CLINICAL TRIAL: NCT06176612
Title: In Patients With Crowe Type III and Crowe Type IV Hip Dysplasia, Mid-Term Lower Extremities and Spine After Total Hip Arthroplasty Natural Course
Brief Title: In Patients With Hip Dysplasia, Mid-Term Lower Extremities and Spine After Hip Arthroplasty Natural Course
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A10207
Record Dates: First submitted 2023-12-10; First posted 2023-12-19 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Total Hip Arthroplasty
Keywords: hip; Total hip arthroplasty; developmental hip dysplasia
MeSH Terms: conditions — Developmental Dysplasia of the Hip | interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with Crowe type 3 or Crowe type 4 hip dysplasia who underwent total hip replacement (Experimental)
  Interventions: Procedure: total hip arthroplasty

INTERVENTIONS:
Procedure: total hip arthroplasty — Patients with Crowe type 3 or Crowe type 4 hip dysplasia who underwent hip replacement

SUMMARY:
Patients with developmental hip dysplasia often present to the outpatient clinic in adulthood with hip pain due to progressive hip osteoarthritis. However, they may have complaints such as limping, lumbar lordosis, lower back pain, and leg length difference. Today, the best treatment option for these patients is hip arthroplasty. Hip arthroplasty causes a high rate of functional improvement and pain relief. According to the hip arthroplasty technique applied, improvement in lameness, leg length difference and spinal curvatures is expected. The aim of our study is to show the change in postoperative spine and lower extremity curvatures after hip arthroplasty in patients with advanced developmental hip dislocation.

DETAILED DESCRIPTION:
Developmental hip dysplasia (DDH) describes the spectrum of anatomical changes in the acetabulum and proximal femur; these can cause limping, lower back pain, lumbar lordosis, and leg length variation. DDH is the main cause of degenerative arthritis of the hip and valgus deformity of the knee. The best treatment option for DDH is total hip arthroplasty (THA). During THA, the distorted anatomy of the acetabulum and proximal femur poses great difficulties. Additionally, the soft tissue can be released and the femur can be shortened while correcting the placement of the acetabulum to prevent neurological damage (sciatic nerve paralysis). Postoperative evaluations focused on assessing joint function and alleviating preoperative clinical symptoms. Some studies have examined changes in lower extremity and knee alignment after THA in patients with DDH. In patients with DDH, THA may cause genu valgus deformity due to increased lower extremity length and Q angle immediately after the operation. THA extends the lower extremity, affecting the patellofemoral joint and anterior knee pain. However, the long-term effects of THA on the alignment of the lower extremity are unclear, especially in patients with Crowe type III and IV DDH, which involves femoral shortening osteotomy. There are few studies examining changes in the knee and lower extremities as a result of THA in patients with DDH. The aim of this study is to evaluate the mid- and long-term alignment of the spine and lower extremity after THA with or without femoral shortening osteotomy in patients with unilateral DDH (Crowe type III-IV).

ELIGIBILITY:
Inclusion Criteria:

1. Patients with unilateral Crowe type 3 hip dysplasia
2. Patients with unilateral Crowe type 4 hip dysplasia

Exclusion Criteria:

1. Patients with unilateral Crowe type 1 hip dysplasia
2. Patients with unilateral Crowe type 2 hip dysplasia
3. History of previous surgery on the hip for which surgery is planned

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2021-04-15 (Actual); Primary Completion 2023-11-15 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Mechanical axis deviation (MAD) | From enrollment to the end of treatment at 2 years
  the lower limb was defined as the distance from the center of the knee to the mechanical axis of the lower limb

SECONDARY OUTCOMES:
tibiofemoral angle (TFA) | From enrollment to the end of treatment at 2 years
  the angle formed by the line from the center of the femoral canal to the center of the knee joint and the line from the center of the knee joint to the center of the ankle joint.
The femoral offset (FO) | From enrollment to the end of treatment at 2 years
  the vertical distances from the center of the femoral head to the center of the femoral canal
The hip-knee-ankle angle (HKA) | From enrollment to the end of treatment at 2 years
  the angle formed by the mechanical axis of the femur and the mechanical axis of the tibia
The lateral distal femoral angle (LDFA) | From enrollment to the end of treatment at 2 years
  the angle formed by the anatomic axis of the femur and the distal femoral joint orientation line
The medial proximal tibial angle (MPTA) | From enrollment to the end of treatment at 2 years
  the angle formed by the anatomic axis of the tibia and the proximal tibial joint orientation line

CONTACTS AND LOCATIONS:
Locations (1):
- Bezmialem Vakıf University, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
I do not think it is right that the data of the patients in the study can be seen by everyone.

REFERENCES:
- [Result] Can A, Erdogan F, Yontar NS, Ovul Erdogan A, Erdem MN, Sarikaya IA. Spinopelvic alignment does not change after bilateral total hip arthroplasty in patients with bilateral Crowe type-IV developmental dysplasia of the hip. Acta Orthop Traumatol Turc. 2020 Nov;54(6):583-586. doi: 10.5152/j.aott.2020.19043. PMID 33423988
- [Result] Zhao HY, Kang PD, Shi XJ, Zhou ZK, Yang J, Shen B, Pei FX. Effects of Total Hip Arthroplasty on Axial Alignment of the Lower Limb in Patients with Unilateral Developmental Hip Dysplasia (Crowe type IV). J Arthroplasty. 2019 Oct;34(10):2406-2414. doi: 10.1016/j.arth.2019.04.028. Epub 2019 Apr 20. PMID 31103361
- [Result] Kocabiyik A, Misir A, Kizkapan TB, Yildiz KI, Kaygusuz MA, Alpay Y, Ezici A. Changes in Hip, Knee, and Ankle Coronal Alignments After Total Hip Arthroplasty With Transverse Femoral Shortening Osteotomy for Unilateral Crowe Type IV Developmental Dysplasia of the Hip. J Arthroplasty. 2017 Nov;32(11):3449-3456. doi: 10.1016/j.arth.2017.05.044. Epub 2017 Jun 1. PMID 28641973